CLINICAL TRIAL: NCT04920422
Title: Dosing Patterns With Regorafenib in Clinical Practice in Spain: A Retrospective Study.
Brief Title: RE-SEARCH Study: A Study to Learn How and in Which Amount Regorafenib is Given in Usual Practice to Patients in Spain: a Study Looking Back at Cases That Have Already Happened When the Study Begins.
Acronym: RE-SEARCH
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21749
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; Refractory metastatic colorectal cancer; Observational Study; Regorafenib
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic colorectal cancer patients.: Medical history data of all patients with at least 1 treatment with regorafenib will be collected retrospectively.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Retrospective analysis using database without any intervention assigned in the study.

SUMMARY:
Researchers are collecting more information to improve treatment of metastatic colorectal cancer (mCRC) with regorafenib.

Metastatic colorectal cancer (mCRC) is a cancer that starts in the large bowel and involves the rectum (the lowest part of the gut) and has spread to other parts of the body. Regorafenib is available to treat patients with mCRC that have previously been treated with, or are not considered candidates for, available therapies. It is an anti-cancer drug that blocks several proteins called enzymes which are involved in the growth of cancer. It is known that doctors may change the amount (the dose) of regorafenib they give, so that the patients better tolerate the treatment. Little information is however available on the doses of regorafenib given in Spain in usual practice.

In this study researchers want to learn how and in which amount regorafenib is usually given to patients with mCRC in Spain. They aim to identify the starting dose of regorafenib and to describe dosing patterns during the first two four-week treatment periods (cycles) according to usual clinical practice.

To answer these questions, the researchers will look back at cases that have already happened when the study begins. Medical history data from the day of diagnosis of the mCRC until the day prior to the inclusion in the study is collected from the medical records of adult patients with mCRC. All patients must have started their treatment with regorafenib since January 2017 and have taken regorafenib for at least 3 months.

The researchers will collect the information between around June 2021 until around November 2021. The final report is planned to be available in July 2022.

No investigational products will be administered in this study. Moreover, no additional visits or laboratory tests will be performed apart from the usual tests/treatments done in usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years
* Patients with histological confirmation of mCRC
* Patient who started treatment with regorafenib for mCRC according to usual clinical practice during or after January 2017 and at least 3 months prior to the inclusion in the study

Exclusion Criteria:

* Patient who have been treated with regorafenib during their participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spanish participants will be included in this study if they had at least one dose of regorafenib in past treatment cycle.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients that start regorafenib treatment with a dose of 80 mg. | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
Percentage of patients that start regorafenib treatment with a dose of 120 mg | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
Percentage of patients that start regorafenib treatment with a dose of 160 mg | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
Percentage of patients that follow each dosing patterns during first two cycles of treatment | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.

SECONDARY OUTCOMES:
Median number of previous lines of treatment received for metastatic colorectal cancer (mCRC) at index. | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  At index (at regorafenib start date)
Percentage of patients according to number of previous lines received at index. | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  At index (at regorafenib start date)
Median time from mCRC diagnosis | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  At index (at regorafenib start date)
Median number of metastatic locations | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  At index (at regorafenib start date)
Percentage of patients with ECOG performance status at index | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  ECOG: Eastern Cooperative Oncology Group.
Percentage of patients with comorbidities at index. | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  At index (at regorafenib start date)
Percentage of patients with mutated BRAF status at index | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  At index (at regorafenib start date)
Percentage of patients with mutated KRAS status at index. | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  At index (at regorafenib start date)
Median duration of regorafenib treatment (cycles) | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  At follow-up
Median progression free survival | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  At follow-up
Percentage of patients for each reason of dose modification. | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.
  At follow-up
Percentage of patients that start cycle 3 based on dosing patterns. | Retrospective data analysis from January 2017 to at least 3 months prior to being included in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Spain

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/